CLINICAL TRIAL: NCT03361020
Title: Obstructive Sleep Apnea in Survivors of Hodgkin Lymphoma Treated With Thoracic Radiation
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: APNEA; R01CA215405 (NIH)
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea; Hodgkin Lymphoma
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hodgkin Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hodgkin Lymphoma: Participants will be survivors of Hodgkin Lymphoma (HL) who were treated with thoracic radiation during the course of their HL, who meet eligibility criteria, and who consent to this study.
- Control Group: The Comparison or control group members will be recruited from healthy parents, sibling, relative or friends who accompany the participant for follow-up at SJCRH and who meet eligibility criteria.

SUMMARY:
While thoracic radiation therapy (TRT) has been a primary component in successful treatment of Hodgkin lymphoma, exposure to this treatment has been associated with significant cardiovascular, cerebrovascular, and pulmonary morbidity in long-term survivors. Survivors of Hodgkin lymphoma (HL) are also at risk for fatigue and excessive daytime sleepiness. Insufficient sleep is recognized as an important public health concern, and is associated with cardiovascular disease, diabetes, obesity, neurocognitive problems, and reduced quality of life and productivity.

Survivors of HL, who are already at risk for cardiac and neurologic morbidity due to their treatment exposures, could face catastrophic cardiovascular and cerebrovascular events with the added risk associated with obstructive sleep apnea (OSA). The investigators propose to examine indices of sleep quality using polysomnography, and associated neurocognitive performance, brain MRI, and structure and strength of neck muscles in 220 long-term adult survivors of Hodgkin lymphoma treated with thoracic radiation.

OBJECTIVES:

1. To estimate the prevalence of OSA in adult survivors of HL treated with thoracic radiation, and compare the frequency to community controls matched on age, gender, race and body mass index.
2. To identify specific therapeutic factors associated with OSA in adult survivors of HL treated with thoracic radiation.
3. To identify biomarkers of OSA in adult survivors of HL treated with thoracic radiation.
4. To examine associations between OSA and cardiac morbidity and brain integrity in the adult survivors of HL treated with thoracic radiation.

DETAILED DESCRIPTION:
Hodgkin lymphoma (HL) survivors being following at St. Jude within the SJLIFE protocol cohort who were treated with TRT will be recruited to complete a comprehensive neurocognitive evaluation, overnight polysomnography evaluation, brain and neck MRI, cervical strength testing, and serum biomarkers related to cardiac disease. As part of their standard SJLIFE evaluation, they will also complete an echocardiogram, pulmonary function tests and questionnaires designed to evaluate broad health, emotional, socioeconomic and environmental factors that impact everyday life.

The investigators will also recruit a comparison sample of healthy individuals matching on age, sex, race and body mass index. The comparison group will complete the comprehensive neurocognitive evaluation, overnight polysomnography, neck MRI, and cervical strength testing.

ELIGIBILITY:
HODGKIN LYMPHOMA SURVIVOR ELIGIBILITY CRITERIA

Inclusion Criteria (Hodgkin Lymphoma Survivor):

* Current participant in the SJLIFE clinical trial ongoing at St. Jude Children's Research Hospital (SJCRH) and was treated with thoracic radiation for Hodgkin lymphoma
* Currently ≥ 18 years of age
* ≥ 5 years from original diagnosis

Exclusion Criteria (Hodgkin Lymphoma Survivor):

* History of cranial or total-body radiation therapy
* History of intrathecal Methotrexate, high-dose Methotrexate, or high-dose Cytarabine.
* History of head injury or diagnosis of a genetic disorder associated with neurocognitive impairment
* History of a neurodevelopmental disorder or birth complication associated with neurocognitive impairment
* History of congenital heart disease reported in the literature to be associated with neurocognitive status as determined by the PIs
* Currently pregnant
* Secondary central nervous system (CNS) neoplasm

COMPARISON GROUP (CONTROL) ELIGIBILITY CRITERIA

Inclusion Criteria (Comparison Group):

* Research participant is a sibling, parent, relative or friend of a current or former St. Jude patient
* Research participant must be at least 18 years of age at the time of the scheduled evaluation

Exclusion Criteria (Comparison Group):

* History of cranial, total-body or thoracic radiation therapy
* History of intrathecal Methotrexate, high-dose Methotrexate, or high-dose Cytarabine.
* History of head injury or diagnosis of a genetic disorder associated with neurocognitive impairment
* History of a neurodevelopmental disorder or birth complication associated with neurocognitive impairment
* History of congenital heart disease reported in the literature to be associated with neurocognitive status as determined by the PIs
* Currently pregnant
* History of cancer
* 1st degree relative of a survivor included in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be survivors of Hodgkin Lymphoma (HL) who were treated with thoracic radiation during the course of their HL, who meet eligibility criteria, and who consent to this study. The Comparison or control group members will be recruited from healthy parents, sibling, relative or friends who accompany the participant for follow-up at SJCRH and who meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 434 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with obstructive sleep apnea (OSA) compared between groups | Once, at enrollment
  The comparison will be between the Hodgkin lymphoma survivors and race, age, sex, body mass index (BMI) matched control group on frequency of OSA. OSA will be deemed present if either of two conditions is met: (1) polysomnography reveals an apnea hypopnea index (AHI) ≥ 15, or (2) polysomnography reveals an AHI ≥ 5 and the participant presents with clinical symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Krull, PhD, Principal Investigator — St. Jude Children's Research Hospital; Belinda Mandrell, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols